CLINICAL TRIAL: NCT00786123
Title: Exploring the Mechanism of a Probiotic Combination VSL#3 in Irritable Bowel Syndrome: a Randomized Double Blind Placebo Controlled Study
Brief Title: Exploring the Mechanism of a Probiotic Combination VSL#3 in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Khek Yu Ho / Professor, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D/06/136
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; rectal hypersensitivity; probiotics; melatonin; brain-gut axis
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 (Experimental): Patients taking probiotics (VSL#3)
  Interventions: Dietary Supplement: VSL#3
- Placebo (Placebo Comparator): Identical looking preparation of placebo taken at the same dose regimen as the active comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — Dose: 4 capsules of VSL#3 daily for 6 weeks.
  Other Names: probiotics
  Arms: VSL#3
Dietary Supplement: Placebo — Identical looking preparation of placebo taken at the same dose regimen as the active comparator
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) is a very common chronic gastrointestinal disorder. Existing therapies for IBS are still far from satisfactory and new therapies are being constantly sought. Probiotics are promising candidate for the prevention and treatment of IBS. However, its efficacy and mechanism is still unclear. The current study aims to evaluate the effects of a combination probiotic, VSL#3, on symptoms and rectal sensitivity in patients with IBS. The underlying mechanism will also be investigated. We will recruit forty patients with Rome III IBS and randomized them, in a parallel group, double-blinded design, to take four VSL#3 capsules or placebos, twice daily, for six weeks. Before and after treatment, patients will be assessed for their symptoms, rectal sensitivity, as well as saliva and fecal melatonin levels. Bowel symptom diary and weekly satisfactory relief of bowel symptoms will also be recorded and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients with IBS between the ages of 18 and 68 will be recruited. IBS will be diagnosed according to the Rome III diagnostic criteria (Drossman and Dumitrascu, 2006). The history of previous chronic GI symptoms suggestive of IBS should be at least 3 months (not necessarily consecutive) over the preceding 6 months. The stool culture of each subject should be negative for hemoccult, pathogens (Salmonella and Shigella), parasites (Giardia) and ova/ cyst. Only patients who had IBS symptoms for at least one month prior to the study and whose IBS symptom score is of at least a moderate severity on at least one of IBS symptoms will be eligible for inclusion into the study.

Exclusion Criteria:

* Those subjects who are unwilling or unable to give informed consent, follow protocol or to stop all medications used to treat diarrhoea or colitis
* Subject taking at the time of proposed enrolment any of the below listed prohibited medications:

  * Anticholinergics (dicyclomine, hyoscyamine, propantheline)
  * Cholinomimetic agents (bethanechol etc.)
  * All narcotics (morphine, codeine, propoxyphene either alone or in any
  * combination)
  * 5-HT3 receptor antagonists (e.g., alosetron, ondansetron, tropisetron, dolasetron, granisetron).
  * Gastrointestinal preparations:
  * Antacids (containing either magnesium or aluminium)
  * Antidiarrheal agents
  * Bismuth compounds
  * Laxatives (stimulant or osmotic)
  * Sulfasalazine
* Treatment with immunosuppressive medications or presence of an immunocompromised state
* If currently using medication (like those used in Diabetes mellitus, Sarcoidosis, Connective tissue disease, poorly controlled hypo/hyperthyroidism) may alter bowel motility or if under long term antibiotic therapy
* Use of any other investigational drug and/or participation in any clinical trial within 3 months of entry to this study
* Patients will be excluded if they had undergone previous abdominal surgery (except appendectomy, Caesarean section, Cholecystectomy, Tubal ligation, Hysterectomy, Hernia repair ≥ 6 months prior to enrolment)
* Subject who has been diagnosed with any of the following GI disorders:

  * Inflammatory bowel disease (Crohn's disease, Ulcerative colitis, Indeterminate Colitis
  * Microscopic colitis (lymphocytic colitis, collagenous colitis)
  * Celiac Disease
  * Gastroparesis
  * Gastrointestinal obstruction and/or stricture
  * Chronic pancreatitis
* Subject with a significant concomitant psychiatric, neurological, metabolic, renal, hepatic, infections, hematological, C.V or pulmonary illness, unless condition is stable and judged by the investigator that such condition does not interfere with the patients participation in the study.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Resolution of symptoms | 6 weeks

SECONDARY OUTCOMES:
Rectal sensitivity | 6 weeks
Saliva and fecal melatonin levels | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ho Khek Yu, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Camilleri M. Is there a role for probiotics in irritable bowel syndrome? Dig Liver Dis. 2006 Dec;38 Suppl 2:S266-9. doi: 10.1016/S1590-8658(07)60007-3. PMID 17259088
- [Background] Shen B, Brzezinski A, Fazio VW, Remzi FH, Achkar JP, Bennett AE, Sherman K, Lashner BA. Maintenance therapy with a probiotic in antibiotic-dependent pouchitis: experience in clinical practice. Aliment Pharmacol Ther. 2005 Oct 15;22(8):721-8. doi: 10.1111/j.1365-2036.2005.02642.x. PMID 16197493
- [Background] Song GH, Venkatraman V, Ho KY, Chee MW, Yeoh KG, Wilder-Smith CH. Cortical effects of anticipation and endogenous modulation of visceral pain assessed by functional brain MRI in irritable bowel syndrome patients and healthy controls. Pain. 2006 Dec 15;126(1-3):79-90. doi: 10.1016/j.pain.2006.06.017. Epub 2006 Jul 18. PMID 16846694
- [Background] Song GH, Leng PH, Gwee KA, Moochhala SM, Ho KY. Melatonin improves abdominal pain in irritable bowel syndrome patients who have sleep disturbances: a randomised, double blind, placebo controlled study. Gut. 2005 Oct;54(10):1402-7. doi: 10.1136/gut.2004.062034. Epub 2005 May 24. PMID 15914575